CLINICAL TRIAL: NCT02174939
Title: Cilostazol Enhances the Number and Functions of Circulating Endothelial Progenitor Cells and Endothelial Function Mediated Through Modification of Vasculogenesis and Angiogenesis Factors in Patients With Stable Coronary Artery Disease
Brief Title: Effect of Cilostazol on Endothelial Progenitor Cells and Endothelial Function in Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-BR-102-076; NCKUH-10304022 (Other Grant/Funding Number: NCKUH)
Record Dates: First submitted 2014-06-22; First posted 2014-06-26 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Disease
Keywords: cilostazol; progenitor cells; coronary artery disease; myocardial infarction; angiogenesis; biological markers; endothelial function
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (Active Comparator): One tablet (100 mg) twice per day for 12 weeks
  Interventions: Drug: Cilostazol
- Dummy Placebo (Placebo Comparator): One tablet twice per day for 12 weeks
  Interventions: Drug: Dummy Placebo

INTERVENTIONS:
Drug: Cilostazol — One tablet (100 mg) twice per day for 12 weeks
  Other Names: Pletaal (brand name)
  Arms: Cilostazol
Drug: Dummy Placebo — One tablet twice per day for 12 weeks
  Other Names: Placebo; Control
  Arms: Dummy Placebo

SUMMARY:
1. The number and function of circulating endothelial progenitor cells (EPCs) are inversely associated with coronary risk factors and atherosclerotic diseases such as coronary artery disease (CAD) and cardiovascular high risk.
2. This double-blind, randomized, placebo-controlled trial to evaluate the effects of cilostazol on human early EPCs and endothelial function as well as the potential mechanisms of action in patients with CAD and cardiovascular high risk.

DETAILED DESCRIPTION:
1. titration of drugs

   1. run-in period: eligible subjects are screened and baseline blood samples are obtained
   2. study period: 12 weeks

      * subjects with cilostazol and subjects with dummy placebo
      * On the first day after the end of the study period, the follow-up data are obtained by the same procedure
   3. blood sampling and measurement of serum biomarkers

      * obtained from peripheral veins in all study subjects at the run-in period and the end of the treatment period of the study
      * sent for isolation, cell culture, and assays of human EPCs
      * also stored for enzyme-linked immunosorbent assay (Stromal cell derived factor-alfa1, adiponectin, soluble thrombomodulin, vascular endothelial growth factor)
2. assays of human EPCs

   1. colony formation by EPCs
   2. quantification of EPCs and apoptotic endothelial cells
   3. chemotactic motility, proliferation/viability and apoptosis assays
3. measurement of flow-mediated dilatation (FMD) of left brachial artery by sonography
4. assessment of long-term cardiovascular outcomes

ELIGIBILITY:
Inclusion Criteria:

* stable CAD documented by stress test, computed tomography angiography or coronary angiography or
* old myocardial infarction (>6 months)
* history and evidence of CAD
* history and evidence of cerebrovascular accident
* history and evidence of peripheral artery disease
* diabetes mellitus
* metabolic syndrome
* stage 3 to 5 chronic kidney disease
* at least 2 of the followings: male ≥45 years old or female ≥55 years old; hypertension; current or past 3-year tobacco smoking; hyperlipidemia; family history of premature CAD (male <55 years old or female <65 years old)

Exclusion Criteria:

* unstable CAD
* have plan to do percutaneous intervention or bypass surgery for CAD or peripheral artery disease within recent 3 months
* severe liver dysfunction (transaminases >10 times of upper normal limit, history of liver cirrhosis, or hepatoma)
* left ventricular ejection fraction (<50% by echocardiography)
* documented active malignancy
* chronic inflammatory disease
* known drug allergy history for cilostazol
* current use of cilostazol or any other cAMP-elevator
* premenopausal women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Circulating EPCs Number | 3 months
  Peripheral blood mononuclear cells (one million cells in each) are suspended in 100 µL phosphate-buffered saline and incubated for 30 min with monoclonal antibodies against human peridinin chlorophyll protein-conjugated cluster of differentiation antigen-45, phycoerythrin-conjugated anti-human cluster of differentiation antigen-34 antibody and anti-human kinase insert domain receptor (KDR) antibody conjugated with Alexa Flour 647. Cells are washed and analyzed on a FACSCalibur flow cytometer with 100,000 events in the lymphocyte gate. EPCs, which are defined as negative for cluster of differentiation antigen-45 and positive for cluster of differentiation antigen-34 and KDR. Based on the peripheral blood mononuclear cell counts, the absolute number of circulating EPCs/µL is calculated.

SECONDARY OUTCOMES:
Viability (Proliferation) of EPCs | 3 months
  250,000 cells are seeded in each well of a 96-well plate and the cells are added with 200 μl of the culture medium and incubated at 37°C. Medium change is performed 3 days later. On 7th day, the plate is then re-incubated with 100 μl fresh medium and additional 50 μl of 2,3-Bis-(2-Methoxy-4-Nitro-5-Sulfophenyl)-2 Hydrogen-Tetrazolium-5-Carboxanilide reagent, and further incubated in dark at 37°C for 4 h. After incubation, the orange colored complex formed is read at 450 nm using a microplate reader with a 450 nm reference filter.
Composite Major Adverse Cardiovascular Events (MACE) | at least 1 year
  This composite endpoint includes cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, congestive heart failure hospitalization, and target vessel revascularization.
composite major coronary events | at least 1 year
  This composite endpoint includes fatal or nonfatal myocardial infarction, recurrent angina pectoris, and target vessel revascularization.

OTHER OUTCOMES:
FMD of the Brachial Artery | 3 months
  FMD in response to reactive hyperemia is measured in the left brachial artery in a quiet, temperature-controlled room after 10 min of bed rest. A high-resolution ultrasound machine equipped with a 7.5 mega Hertz linear array probe is used for the study. Arterial diameters are measured at the baseline and during reactive hyperemia. FMD is calculated as the percentage change in diameter compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Hsing Chao, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Background] Chao TH, Tseng SY, Li YH, Liu PY, Cho CL, Shi GY, Wu HL, Chen JH. A novel vasculo-angiogenic effect of cilostazol mediated by cross-talk between multiple signalling pathways including the ERK/p38 MAPK signalling transduction cascade. Clin Sci (Lond). 2012 Aug 1;123(3):147-59. doi: 10.1042/CS20110432. PMID 22339730
- [Background] Biscetti F, Pecorini G, Straface G, Arena V, Stigliano E, Rutella S, Locatelli F, Angelini F, Ghirlanda G, Flex A. Cilostazol promotes angiogenesis after peripheral ischemia through a VEGF-dependent mechanism. Int J Cardiol. 2013 Aug 10;167(3):910-6. doi: 10.1016/j.ijcard.2012.03.103. Epub 2012 Apr 2. PMID 22473072
- [Background] Chao TH, Tseng SY, Chen IC, Tsai YS, Huang YY, Liu PY, Ou HY, Li YH, Wu HL, Cho CL, Tsai LM, Chen JH. Cilostazol enhances mobilization and proliferation of endothelial progenitor cells and collateral formation by modifying vasculo-angiogenic biomarkers in peripheral arterial disease. Int J Cardiol. 2014 Mar 15;172(2):e371-4. doi: 10.1016/j.ijcard.2013.12.295. Epub 2014 Jan 11. No abstract available. PMID 24439864